CLINICAL TRIAL: NCT00976963
Title: Single Dose Monurol for Treatment of Acute Cystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Ann Stapleton, Professor, Medicine, Infectious Diseases, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34776
Record Dates: First submitted 2009-09-11; First posted 2009-09-15 (Estimated); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Urinary Tract Infection
Keywords: UTI
MeSH Terms: conditions — Urinary Tract Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Fosfomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMP/SMX (Active Comparator): Sulfamethoxazole-Trimethoprim 800-160 MG Oral Tab; 800mg/160mg BID x 3 days
  Interventions: Drug: TMP/SMX
- Fosfomycin (Experimental): 3g sachet single dose
  Interventions: Drug: Fosfomycin

INTERVENTIONS:
Drug: TMP/SMX — Take one twice daily for 3 days for urinary tract infection
  Other Names: Septra; Bactrim
  Arms: TMP/SMX
Drug: Fosfomycin — Mix sachet with 1/2 glass cold water and stir. Drink immediately
  Other Names: Monurol
  Arms: Fosfomycin

SUMMARY:
Urinary tract infecton (UTI) is a very common problem in young healthy women, afflicting approximately one-half of women by their late 20's. One of the most common antibiotics used to treat UTIs is Trimethoprim-Sulfamethoxazole (TMP-SMX), usually for total of three days. However, concerns about increased antibiotic resistance have led to increased interest in studying other antibiotics for UTI.

An alternative antibiotic which is also FDA approved for the treatment of UTIs is fosfomycin (Monurol). The effectiveness of fosfomycin in curing UTIs when given as a single dose is not well studied. The purpose of this research study is to determine what the cure rates are with a single dose of fosfomycin versus the more standard 3-day course of TMP-SMX.

DETAILED DESCRIPTION:
Procedures subjects will undergo once they have read and signed the consent are:

Questions about their medical and sexual history and current symptoms of UTI. They will be asked to provide a urine and peri-urethral sample and then are randomly assigned to one of the two treatment groups.They will be given a sheet to record symptoms at home. They will be asked to return to the clinic in 5-8 and 28-30 days after completing antibiotic therapy.Follow-up questions will be asked and urine and peri-urethral will be self collected at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant women in good health with symptoms of acute cystitis for less than 7 days

Exclusion Criteria:

* Pregnant, lactating, or not regularly contracepting
* History of chronic conditions such as diabetes
* Known anatomic abnormalities of the urinary tract
* Use of prophylactic antibiotics
* History of allergy or intolerance to any of the study drugs
* Recent (> 2 weeks)exposure to oral or parenteral antimicrobial
* History of UTI in previous 1 month

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2009-09-17 (Actual); Primary Completion 2016-12-27 (Actual); Study Completion 2016-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann E. Stapleton, M.D., Principal Investigator — University of WA
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women presenting with symptoms of acute uncomplicated cystitis (AUC) at the University of Washington health center were screened for eligibility between September, 2009 to November, 2016
Pre-assignment Details: Of 508 AUC presenters assessed, 208 were excluded due to not meeting inclusion criteria, refusal to participate, or other reasons. 300 were enrolled and randomized to treatment intervention.
Groups:
- TMP/SMX: Sulfamethoxazole-Trimethoprim 800-160 MG Oral Tab; 160/800mg BID x 3 days
  TMP/SMX : Take one twice daily for 3 days for urinary tract infection
Period: Overall Study
Arm/Group | TMP/SMX | Fosfomycin
Started | 150 | 150
Treated With Assigned Intervention | 146 (Participants who were not treated with the assigned randomization therapy were excluded from the main efficacy analyses, "Cure".) | 150
Completed | 146 | 150
Not Completed | 4 | 0
Not completed — medication not dispensed at the pharmacy due to contraindications to the assigned therapy | 2 | 0
Not completed — administrative error | 1 | 0
Not completed — allergic reaction due to previously unknown allergy | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who were dispensed the treatment intervention, completed some or all of the treatment intervention and were included in the summary of side effects.
Groups:
- Total: Total of all reporting groups
Arm/Group | TMP/SMX | Fosfomycin | Total
Number analyzed (Participants) | 147 | 150 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (3) | 21 (3) | 21 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 150 | 297
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 18 | 25
  Not Hispanic or Latino | 140 | 132 | 272
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 90 | 95 | 185
  Asian or Pacific Islander | 39 | 38 | 77
  Other | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Cured
Description: Cure as defined by no further treatment for subsequent or unresolved symptoms, by modified ITT approach.
Time Frame: 28-30 days post therapy
Measure: Count of Participants; unit: Participants
Arm/Group | TMP/SMX | Fosfomycin
Number analyzed (Participants) | 146 | 150
Participants | 120 | 130
Statistical Analysis 1: Comparison: TMP/SMX vs Fosfomycin; The null hypothesis is that Fosfomycin is inferior to TMP/SMX; Test type: Non-Inferiority — The equivalence margin for non-inferiority of Fosfomycin to TMP/SMX is 10%; p < 0.001, Wald test for noninferiority

ADVERSE EVENTS:
Time Frame: 30 days
Description: All participants enrolled (N = 150 in each arm) were monitored for mortality or serious adverse events due to inherent processes in the campus health care system.
  Other adverse events were collected at the 1st follow-up visit in participants who presented for this visit, and they were queried on each side effect.
Arm/Group | TMP/SMX | Fosfomycin
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 46/143 | 43/145
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMP/SMX (N=143) | Fosfomycin (N=145)
Nausea (Gastrointestinal disorders) | 22 | 3
Loose stools (Gastrointestinal disorders) | 7 | 28
Abdominal discomfort (Gastrointestinal disorders) | 10 | 12
Headache (General disorders) | 11 | 3
Dizziness (General disorders) | 7 | 3
Fatigue/weakness (General disorders) | 8 | 6

LIMITATIONS AND CAVEATS:
The clinicians and participants were not blinded as to the assigned intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No